CLINICAL TRIAL: NCT00281892
Title: Darbepoetin Alfa in Patients With Chronic Lymphocytic Leukemia and Comorbidity
Brief Title: Fludarabine and Darbepoetin Alfa in Treating Older Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL9; GCLLSG-CLL9; EU-20561; AMGEN-GCLLSG-CLL9; 2005-003014-15 (EudraCT Number)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Chronic Lymphocytic Leukemia; Anemia
Keywords: anemia; refractory chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Anemia | interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fludarabine plus Darbopoetin (Experimental): Group 1 - Patients with an initial Hb-value of less than 12 g/dl receive fludarabine (30 mg/m² intravenously on day 1, 3, 5; repeated every 28 days for 6 cycles and 500 mcg of darbepoetin alfa subcutaneously every 3 weeks
  Interventions: Biological: Fludarabine plus Darbopoetin
- fludarabine mono (Active Comparator): Group 1 - Patients with an initial Hb-value of less than 12 g/dl receive fludarabine (30 mg/m² intravenously on day 1, 3, 5; repeated every 28 days for 6 cycles with no additional growth factor support.
  Group 2 - Patients with an initial Hb-value more than 12 g/dl start to receive fludarabine (30 mg/m² intravenously on day 1, 3, 5; repeated every 28 days for 6 cycles . Patients of group 2 will be eventually randomized at later timepoints, if the Hb-value drops below 12 g/dl. Randomized patients will receive either 500 mcg darbepoetin alfa subcutaneously every 3 weeks or continue therapy with fludarabine without additional administration of darbepoetin alfa.
  Interventions: Drug: Fludarabine mono

INTERVENTIONS:
Biological: Fludarabine plus Darbopoetin — Group 1 - Patients with an initial Hb-value of less than 12 g/dl receive fludarabine (30 mg/m² intravenously on day 1, 3, 5; repeated every 28 days for 6 cycles and 500 mcg of darbepoetin alfa subcutaneously every 3 weeks
  Arms: Fludarabine plus Darbopoetin
Drug: Fludarabine mono — Group 1 - Patients with an initial Hb-value of less than 12 g/dl receive fludarabine (30 mg/m² intravenously on day 1, 3, 5; repeated every 28 days for 6 cycles with no additional growth factor support.
  Group 2 - Patients with an initial Hb-value more than 12 g/dl start to receive fludarabine (30 mg/m² intravenously on day 1, 3, 5; repeated every 28 days for 6 cycles . Patients of group 2 will be eventually randomized at later timepoints, if the Hb-value drops below 12 g/dl. Randomized patients will receive either 500 mcg darbepoetin alfa subcutaneously every 3 weeks or continue therapy with fludarabine without additional administration of darbepoetin alfa.
  Arms: fludarabine mono

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Darbepoetin alfa may cause the body to make more red blood cells. It is not yet known whether fludarabine is more effective with or without darbepoetin alfa in treating chronic lymphocytic leukemia.

PURPOSE: This phase III trial is studying fludarabine to see how well it works when given together with or without darbepoetin alfa in treating older patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of fludarabine with or without darbepoetin alfa in geriatric patients with chronic lymphocytic leukemia and relevant comorbidities.
* Determine the effect of these regimens in reducing anemia, lowering the requirements of transfusion, and reducing the duration and frequency of hospitalization in these patients.
* Determine the quality of life of patients treated with these regimens.
* Determine event-free, progression-free, and overall survival of patients treated with these regimens.
* Evaluate the medical-economical aspects of these regimens in these patients

OUTLINE: This is a multicenter study. Patients are stratified according to hemoglobin value (< 12 g/dL [stratum 1] vs > 12 g/dL [stratum 2]). Patients are assigned to 1 of 2 treatment strata.

* Stratum 1: Patients receive fludarabine IV on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses. Patients also receive darbepoetin alfa subcutaneously once weekly for up to 6 weeks.
* Stratum 2: Patients receive fludarabine as in stratum 1. Quality of life is evaluated periodically.

PROJECTED ACCRUAL: A total of 348 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL) meeting 1 of the following criteria:

  * Previously untreated disease
  * Progressive or relapsed CLL after treatment with nonpurine analog-containing regimens as chlorambucil or bendamustine hydrochloride
* Meets 1 of the following staging criteria:

  * Binet stage A disease with B symptoms requiring treatment
  * Binet stage B disease requiring treatment, meeting ≥ 1 of the following criteria:

    * Rapid disease progression
    * Enlarged lymph nodes and organs
    * Severe B symptoms
  * Binet stage C disease
* Must have comorbidities (i.e., CIRS score > 6)
* Must have restricted kidney function (i.e., creatinine clearance < 70mL/min)
* No transformation to aggressive non-Hodgkin's lymphoma (Richter's syndrome)

PATIENT CHARACTERISTICS:

* Life expectancy > 6 months
* Creatinine clearance > 30 mL/min
* No active second malignancy
* No active bacterial, viral, or fungal infection
* No conditions that would preclude substitution of iron
* No severe myocardial, coronary, or respiratory insufficiency
* No severe liver insufficiency
* No known hypersensitivity to darbepoetin alfa
* No cerebral dysfunction that would preclude participation in the required study procedures

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent participation in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2004-09; Primary Completion 2008-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Event-free survival | up to 24 months after the last dose of study medication
  defined as the time from initial randomization/stratification to the time-point of progressive disease, new therapy, or death)

SECONDARY OUTCOMES:
Response Rate | 2 months after the end of the last cycle
  Restaging after the end of treatment included evaluation of the peripheral blood and physical examination; use of imaging techniques (ultrasound and conventional radiography or computertomography) and evaluation of the bone marrow were mandatory to assign a complete remission
toxicity | 28 days after the end of the last cycle
  adverse events were reported according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC version 2.0).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (46):
- Germany (46):
  - Hamatologische/Onkologische Gemeinschaftspraxis - Augsburg, Augsburg
  - Onkologische Schwerpunktpraxis und Tagesklinik Dres, Bad Soden
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Internistische Praxis - Dusseldorf, Düsseldorf
  - Hans - Susemihl - Krankenhaus, Emden
  - Universitaetsklinikum Essen, Essen
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Internistische Praxis - Gerlingen, Gerlingen
  - Internistische Praxisgemeinschaft, Germering
  - Universitaetsklinikum Göttingen, Göttingen
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Kempten Oberallgaeu, Kempten
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Caritas - Krakenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Staedtisches Klinikum Magdeburg, Magdeburg
  - Hospital Maria-Hilf II, Mönchengladbach
  - Munich Oncologic Practice at Elisenhof, Munich
  - I. Frauenklinik und Hebammenschule der Ludwig-Maximillians Universitaet Muenchen, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Haematologische Schwerpunktpraxis, Munich
  - Klinikum Schwaebisch Gmuend Stauferklinik, Mutlangen
  - Hamatologie/Onkologie Praxisgemeinschaft - Muenchen, München
  - Haematologische-onkologische GemeinschaftspraxisSchick - Schick - Schmidt - Wiesmeier, München
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Pforzheim
  - Scherpunktpraxis fur Hematologie und Onkologie, Regensburg
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbrücken
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - St. Marienhospital - Vechta, Vechta
  - Haematologische Praxis, Weiden
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goede V, Busch R, Bahlo J, Chataline V, Kremers S, Muller L, Reschke D, Schlag R, Schmidt B, Vehling-Kaiser U, Wedding U, Stilgenbauer S, Hallek M. Low-dose fludarabine with or without darbepoetin alfa in patients with chronic lymphocytic leukemia and comorbidity: primary results of the CLL9 trial of the German CLL Study Group. Leuk Lymphoma. 2016;57(3):596-603. doi: 10.3109/10428194.2015.1079314. Epub 2015 Oct 12. PMID 26293380
- [Result] Goede V, Bahlo J, Chataline V, Eichhorst B, Durig J, Stilgenbauer S, Kolb G, Honecker F, Wedding U, Hallek M. Evaluation of geriatric assessment in patients with chronic lymphocytic leukemia: Results of the CLL9 trial of the German CLL study group. Leuk Lymphoma. 2016;57(4):789-96. doi: 10.3109/10428194.2015.1091933. Epub 2015 Oct 13. PMID 26377031